CLINICAL TRIAL: NCT00006226
Title: A Phase II Trial of Thalidomide in Patients With Relapsed Chronic Lymphocytic Leukemia
Brief Title: Thalidomide in Treating Patients With Relapsed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01852; NCI-2012-01852 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N9986; CDR0000068148; N9986 (Other: North Central Cancer Treatment Group); N9986 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Thalidomide

ARMS (1):
- Treatment (thalidomide) (Experimental): Patients receive oral thalidomide daily for 4 weeks. Courses repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: thalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: thalidomide — Given PO
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of thalidomide in treating patients who have relapsed chronic lymphocytic leukemia. Thalidomide may stop the growth of chronic lymphocytic leukemia by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether thalidomide can induce objective responses in relapsed B-CLL patients.

II. To determine the toxicity of thalidomide in this patient population. III. To document if alterations in vascular growth factors and/or bone marrow angiogenesis patterns correlate with thalidomide related clinical responses.

OUTLINE:

Patients receive oral thalidomide daily for 4 weeks. Courses repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) evidenced by monoclonal population of mature CD5+, CD19+, CD23+, and B cells
* Relapsed after prior treatment for CLL
* Active disease with 1 or more of the following characteristics:

  * At least 10% weight loss within the past 6 months
  * Fever greater than 100.5 degrees F for at least 2 weeks without evidence of infection
  * Night sweats without evidence of infection
  * Evidence of progressive marrow failure with anemia (hemoglobin less than 11 g/dL) and/or thrombocytopenia (platelet count less than 100,000/mm^3) (i.e., any stage III or IV disease)
  * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy
  * Massive or progressive splenomegaly (i.e., greater than 6 cm below the left costal margin or more than 50% increase over 2 months)
  * Progressive lymphadenopathy (i.e., more than 50% increase over 2 months)
  * Progressive lymphocytosis (not due to corticosteroids) with an increase of more than 50% over a 2-month period or an anticipated doubling time of less than 6 months
  * Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease are not considered evidence of active disease
* Measurable disease

  * Absolute lymphocyte count greater than 5,000/mm^3
* No bulky lymph node disease greater than 10 cm in at least 1 dimension except splenomegaly
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 500/mm^3
* Platelet count at least 20,000/mm^3 (in absence of sargramostim [GM-CSF])
* Hemoglobin at least 8 g/dL
* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No other active malignancy
* No peripheral neuropathy (sensory) grade 2 or greater
* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 1 highly effective method of contraception AND 1 additional effective method of contraception for at least 4 weeks before, during, and for 4 weeks after study completion
* No prior allogeneic bone marrow transplantation
* At least 10 days since prior filgrastim (G-CSF) or GM-CSF
* No more than 3 prior chemotherapy regimens
* At least 30 days since prior chemotherapy
* No concurrent corticosteroids except for adrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2000-09; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Confirmed response, noted as the objective status of CR, nPR, or PR on 2 consecutive evaluations at least 4 weeks apart | Up to 5 years
  Ninety percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  The Kaplan-Meier method will be used.
Progression-free survival | Up to 5 years
  The Kaplan-Meier method will be used.
Time to progression | Up to 5 years
  The Kaplan-Meier method will be used.
Duration of response | Up to 5 years
Maximum grade of each type of toxicity | Up to 5 years
  Frequency tables will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Kay, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States